CLINICAL TRIAL: NCT02676466
Title: The ENRGISE (ENabling Reduction of Low-Grade Inflammation in SEniors) Pilot Study
Acronym: ENRGISE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB201500894 - A-N; U01AG050499 (NIH)
Record Dates: First submitted 2016-02-03; First posted 2016-02-08 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2019-12

CONDITIONS: Inflammation
Keywords: Mobility
MeSH Terms: conditions — Inflammation | interventions — Fish Oils; Losartan; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Fish oil Active (Experimental): This group will receive the Omega-3 fish oil which will be administered at a dose of 1.4 grams per day for the first six months. Based on tolerability and inflammation level, dose may either continue at 1.4 grams per day or be increased to 2.8 grams per day for the remaining six month.
  Interventions: Dietary Supplement: Omega-3 fish oil
- Fish oil Placebo (Placebo Comparator): This group will receive a placebo which will be matching to the Omega-3 fish oil. The placebo corn oil are obtained in gel caps and they have identical shape, color, taste and weight. The doses will be administered at doses corresponding to the Omega-3 fish oil.
  Interventions: Other: Corn Oil (Fish oil Placebo)
- Losartan Active (Active Comparator): This group will receive the Losartan which will be administered at a starting dose of 25 milligrams per day. Based on tolerability, losartan will continue at a dose of either 25 milligrams per day or 50 milligrams per day for the first six months. Based on continued tolerability and inflammation level, dose may either continue at 25 or 50 milligrams per day or be increased to 100 milligrams per day for the remaining six months.
  Interventions: Drug: Losartan
- Losartan Placebo (Placebo Comparator): This group will receive a placebo which will be matching to the losartan. The placebo cellulose based capsule are obtained in 25 mg and 50 mg capsules. The shell capsules are cellulose based. Placebo and LO have identical shape, color, taste and weight. the doses will be administered at doses corresponding to the losartan.
  Interventions: Other: Cellulose Based (Losartan Placebo)
- Fish oil Active + Losartan Active (Active Comparator): This group will receive both the Losartan and Omega-3 fish oil. Losartan will be administered at a starting dose of 25 milligrams per day. Based on tolerability, losartan will continue at a dose of either 25 milligrams per day or 50 milligrams per day for the first six months. Based on continued tolerability and inflammation level, dose may either continue at 25 or 50 milligrams per day or be increased to 100 milligrams per day for the remaining six months.
  Omega-3 fish oil will be administered at a dose of 1.4 grams per day for the first six months. Based on tolerability and inflammation level, dose may either continue at 1.4 grams per day or be increased to 2.8 grams per day for the remaining six month.
  Interventions: Dietary Supplement: Omega-3 fish oil; Drug: Losartan
- Fish oil Active + Losartan Placebo (Other): This group will receive the Omega-3 fish oil which will be administered at a dose of 1.4 grams per day for the first six months. Based on tolerability and inflammation level, dose may either continue at 1.4 grams per day or be increased to 2.8 grams per day for the remaining six month.
  In addition, this group will receive a placebo which will be matching to the losartan. The placebo cellulose based capsule are obtained in 25 mg and 50 mg capsules. The shell capsules are cellulose based. Placebo and LO have identical shape, color, taste and weight. the doses will be administered at doses corresponding to the losartan.
  Interventions: Dietary Supplement: Omega-3 fish oil; Other: Cellulose Based (Losartan Placebo)
- Fish oil Placebo + Losartan Active (Other): This group will receive a placebo which will be matching to the Omega-3 fish oil. The placebo corn oil are obtained in gel caps and they have identical shape, color, taste and weight. The doses will be administered at doses corresponding to the Omega-3 fish oil.
  In addition, this group will receive the Losartan which will be administered at a starting dose of 25 milligrams per day. Based on tolerability, losartan will continue at a dose of either 25 milligrams per day or 50 milligrams per day for the first six months. Based on continued tolerability and inflammation level, dose may either continue at 25 or 50 milligrams per day or be increased to 100 milligrams per day for the remaining six months.
  Interventions: Drug: Losartan; Other: Corn Oil (Fish oil Placebo)
- Fish oil Placebo + Losartan Placebo (Other): This group will receive a placebo which will be matching to both the omega-3 fish oil and losartan which will be administered at doses corresponding to doses administered for omega-3 fish oil and losartan throughout the 12 month study.
  Interventions: Other: Corn Oil (Fish oil Placebo); Other: Cellulose Based (Losartan Placebo)

INTERVENTIONS:
Dietary Supplement: Omega-3 fish oil — The Omega-3 fish oil will be provided in 700 mg gelcaps. The starting dose will be 1.4 g/day of fish oil and continue until the 6 month visit. If the average of IL-6 measured at 3- and 6-month visits does not decrease by >40% vs. baseline (average of screening visits 1 and 2), we increase the dose to 2.8 g/day.
  Arms: Fish oil Active; Fish oil Active + Losartan Active; Fish oil Active + Losartan Placebo
Drug: Losartan — The Losartan will be provided in 25 mg and 50 mg capsules. The starting dose will be 25 mg/day, if tolerated, then stepped up to 50 mg/day. If there are no safety concerns, a continuation of 50 mg/day will be provided until the 6 month visit. If the average of IL-6 measured at 3- and 6-month visits does not decrease by >40% vs. baseline (average of screening visits 1 and 2), an increase to the dose of 100 mg/day.
  Other Names: Cozaar
  Arms: Fish oil Active + Losartan Active; Fish oil Placebo + Losartan Active; Losartan Active
Other: Corn Oil (Fish oil Placebo) — The corn oil placebo gel caps will be identical in shape, color, taste and weight as the Omega-3 fish oil.
  Other Names: Fish oil Placebo
  Arms: Fish oil Placebo; Fish oil Placebo + Losartan Active; Fish oil Placebo + Losartan Placebo
Other: Cellulose Based (Losartan Placebo) — The placebo cellulose based capsules will be identical in shape, color, taste and weight as the losartan capsules.
  Other Names: Losartan Placebo
  Arms: Fish oil Active + Losartan Placebo; Fish oil Placebo + Losartan Placebo; Losartan Placebo

SUMMARY:
ENRGISE Pilot Study will test the ability of anti-inflammatory interventions for preventing major mobility disability by improving or preserving walking ability.

DETAILED DESCRIPTION:
Growing evidence shows that low-grade chronic inflammation, characterized by elevations in plasma C-reactive protein, tumor necrosis factor alpha, and particularly Interleukin-6 (IL-6), is an independent risk factor of disability, impaired mobility, and lower walking speed. Low-grade chronic inflammation is a modifiable risk factor. However, it is unknown whether interventions that reduce the levels of inflammatory markers per se improve mobility, or avert decline in mobility in older persons.

To address this gap in evidence the investigators are conducting the randomized clinical trial ENRGISE (ENabling Reduction of low-Grade Inflammation in SEniors) Pilot Study to test the ability of anti-inflammatory interventions for preventing major mobility disability by improving or preserving walking ability. We have maximized the public health impact by selecting interventions that are safe, tolerable, acceptable, and affordable for vulnerable older persons. Specifically, in this trial the investigators test the efficacy verus placebo of the angiotensin receptor blocker losartan and omega-3 polyunsaturated fatty acids in the form of fish oil, alone and in combination. Both angiotensin receptor blockers and omega-3 polyunsaturated fatty acids have shown to reduce IL-6 in clinical trials and preliminary data suggest that they may improve physical function.

Recruitment will include the older persons who are at risk for, or with, mobility impairment, as measured by slow gait speed and self-reported mobility difficulty, and who have elevated levels of IL-6, the marker most consistently associated with mobility limitations. Preliminary data regarding feasibility need to be gathered before such a trial can be effectively designed and implemented. We conduct The ENRGISE Pilot Study to assess the effects of the interventions on several inflammatory markers, walking speed, physical function and strength. This allows us to refine the design, recruitment yields, target population, adherence, retention, tolerability, sample-size, and cost for the main ENRGISE trial.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age >70 years
* Self-reported difficulty walking ¼ of a mile or climbing a flight of stairs
* Walking speed <1 meters per second and >0.44 meters per second on the 4 meter walk at usual pace. A walking speed of <0.44 meters per second would not be compatible with completing the 400 meter walk in 15 minutes. (In the pilot phase we explore the feasibility of recruiting at least 50% of participants who have a baseline walking speed of <0.80 meters per second and >0.44 meters per second)
* Able to complete the 400 meter walk test within 15 minutes without sitting or the help of another person and without a walker, a cane is allowed
* Blood level IL-6 >2.5 pg/ml and <30 pg/ml.
* Willingness to be randomized to the intervention groups

Exclusion Criteria:

* Failure or inability to provide informed consent
* Lives in a nursing home; persons living in assisted or independent housing are not excluded
* Self-reported inability to walk one block
* Significant cognitive impairment, defined as a known diagnosis of dementia, or a Mini-Mental State Exam (MMSE) score <24 (<23 for racial/ethnic minorities or participants with less than 9 years of education)
* Unable to communicate because of severe hearing loss or speech disorder
* Neurological conditions that are causing impaired muscle function or mobility (may include stroke with residual paresis, paralysis, neuropathy, Parkinson disease, or multiple sclerosis)
* Severe rheumatologic or orthopedic diseases, e.g., awaiting joint replacement, known active inflammatory or autoimmune disease (e.g. rheumatoid arthritis, lupus, Crohn's disease, HIV)
* Terminal illness with life expectancy less than 12 months
* Severe pulmonary disease, requiring either steroid pills or injections
* Other significant co-morbid disease that in the opinion of the field center PI would impair ability to participate in the trial, e.g. renal failure on hemodialysis, severe psychiatric disorder (e.g. bipolar, schizophrenia), excessive alcohol use (>14 drinks per week); drug addiction; treatment for cancer (radiation or chemotherapy) within the past 1 year; or other conditions
* Lives outside of the study site or is planning to move out of the area in next 1 year or leave the area for >3 months during the next year
* Exclusion criteria that apply only to those who receive losartan:

  * Intolerance or allergy to Angiotensin II Receptor Blockers (ARBs)
  * Known bilateral renal artery stenosis or liver cirrhosis
  * Hypotension Systolic Blood Pressure<110 or Diastolic Blood Pressure<60 mmHg
  * Serum potassium ≥5.0 mEq/L
  * Use of lithium salts
  * eGFR <15
  * Congestive heart failure with ejection fraction < 40%
* Exclusion criteria that apply only to those who receive ω-3:

  * Intolerance or allergy to ω-3 or fish/shellfish
  * Fatty fish intake >2 servings per week on average
  * History of paroxysmal or persistent atrial fibrillation
* To maintain blinding, those who are not eligible to receive any active treatment (ω-3 or losartan) are excluded

Temporary exclusion criteria

* Myocardial infarction, coronary artery bypass grafting (CABG), or valve replacement within past 6 months;
* Pulmonary embolism or deep venous thrombosis within past 6 months;
* Uncontrolled diabetes with recent weight loss, diabetic coma, or frequent insulin reactions;
* Stroke, hip fracture, hip or knee replacement, or spinal surgery within past 4 months;
* Physical therapy for gait, balance, or other lower extremity training within the past 2 months;
* Severe hypertension, e.g., Systolic Blood Pressure > 200, or Diastolic Blood Pressure> 110 mmHg;
* Hemoglobin <10 g/dL
* Participation in another intervention trial within 3 months; participation in an observational study may be permitted;
* Current smoking (within 6 months),
* Acute infection (urinary, respiratory, other) or hospitalization within 1 month
* Exclusion criteria that apply only to those who receive losartan:

  * Use of Angiotensin-Converting Enzyme Inhibitor (ACEI), Angiotensin II Receptor Blocker (ARB) within 2 months
  * Use of aliskiren within 2 months in patients with type 2 diabetes or renal impairment with Estimated Glomerular Filtration Rate (eGFR)<60
  * Use of potassium sparing diuretics, other medications with potassium sparing properties (such as but not limited to spironolactone or eplerenone) potassium supplements, and salt substitutes containing potassium within 1 week
  * Transaminases >twice upper limit of normal to exclude participants with impaired liver function
* Exclusion criteria that apply only to those who receive ω-3:

  * Use of ω-3 within 2 months

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 289 (Actual)
Dates: Start 2016-04-26 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Pahor, MD, Principal Investigator — University of Florida; Walter Ambrosius, PhD, Principal Investigator — Wake Forest University
Locations (5):
- United States (5):
  - University of Florida, Gainesville, Florida
  - Northwestern University, Chicago, Illinois
  - Tufts University, Boston, Massachusetts
  - Wake Forest University, Winston-Salem, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The investigator will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for ENRGISE study approved research purposes and not to identify any individual human participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.
Supporting Information: Study Protocol, ICF
Time Frame: per NIH
Access Criteria: per NIH

REFERENCES:
- [Background] Manini TM, Anton SD, Beavers DP, Cauley JA, Espeland MA, Fielding RA, Kritchevsky SB, Leeuwenburgh C, Lewis KH, Liu C, McDermott MM, Miller ME, Tracy RP, Walston JD, Radziszewska B, Lu J, Stowe C, Wu S, Newman AB, Ambrosius WT, Pahor M; ENRGISE Pilot study investigators. ENabling Reduction of Low-grade Inflammation in SEniors Pilot Study: Concept, Rationale, and Design. J Am Geriatr Soc. 2017 Sep;65(9):1961-1968. doi: 10.1111/jgs.14965. Epub 2017 Jul 22. PMID 28734043
- [Derived] Pahor M, Anton SD, Beavers DP, Cauley JA, Fielding RA, Kritchevsky SB, Leeuwenburgh C, Lewis KH, Liu CK, Lovato LC, Lu J, Manini TM, McDermott MM, Miller ME, Newman AB, Radziszewska B, Stowe CL, Tracy RP, Walkup MP, Wu SS, Ambrosius WT. Effect of Losartan and Fish Oil on Plasma IL-6 and Mobility in Older Persons. The ENRGISE Pilot Randomized Clinical Trial. J Gerontol A Biol Sci Med Sci. 2019 Sep 15;74(10):1612-1619. doi: 10.1093/gerona/gly277. PMID 30541065

RESULTS

PARTICIPANT FLOW:
Groups:
- Fish Oil Active + Losartan Active: This group will receive both the Losartan and Omega-3 fish oil. Losartan will be administered at a starting dose of 25 milligrams per day. Based on tolerability, losartan will continue at a dose of either 25 milligrams per day or 50 milligrams per day for the first six months. Based on continued tolerability and inflammation level, dose may either continue at 25 or 50 milligrams per day or be increased to 100 milligrams per day for the remaining six months.
  Omega-3 fish oil will be administered at a dose of 1.4 grams per day for the first six months. Based on tolerability and inflammation level, dose may either continue at 1.4 grams per day or be increased to 2.8 grams per day for the remaining six months.
Period: Overall Study
Arm/Group | Fish Oil Active | Fish Oil Placebo | Losartan Active | Losartan Placebo | Fish Oil Active + Losartan Active | Fish Oil Active + Losartan Placebo | Fish Oil Placebo + Losartan Active | Fish Oil Placebo + Losartan Placebo
Started | 109 | 71 | 26 | 17 | 26 | 13 | 13 | 14
Completed (Recruitment was completed June 22, 2017 and follow-up completed June 22, 2018 in all cells.) | 105 | 66 | 24 | 17 | 23 | 12 | 12 | 13
Not Completed | 4 | 5 | 2 | 0 | 3 | 1 | 1 | 1
Not completed — Death | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 3 | 1 | 0 | 3 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: the baseline analysis population is the same as the analysis population. This is an intent to treat analysis
Groups:
- Fish Oil Active + Losartan Active: This group will receive both the Losartan and Omega-3 fish oil. Losartan will be administered at a starting dose of 25 milligrams per day. Based on tolerability, losartan will continue at a dose of either 25 milligrams per day or 50 milligrams per day for the first six months. Based on continued tolerability and inflammation level, dose may either continue at 25 or 50 milligrams per day or be increased to 100 milligrams per day for the remaining six months.
  Omega-3 fish oil will be administered at a dose of 1.4 grams per day for the first six months. Based on tolerability and inflammation level, dose may either continue at 1.4 grams per day or be increased to 2.8 grams/day for the remaining six month.
  Omega-3 fish oil: The Omega-3 fish oil will be provided in 700 mg gelcaps. The starting dose will be 1.4 g/day of fish oil and continue until the 6 month visit. If the average of IL-6 measured at 3- and 6-month visits does not decrease by >40% vs. baseline (average of screenin
- Fish Oil Active + Losartan Placebo: This group will receive the Omega-3 fish oil which will be administered at a dose of 1.4 grams per day for the first six months. Based on tolerability and inflammation level, dose may either continue at 1.4 grams per day or be increased to 2.8 grams/day for the remaining six month.
  In addition, this group will receive a placebo which will be matching to the losartan. The placebo cellulose based capsule are obtained in 25 mg and 50 mg capsules. The shell capsules are cellulose based. Placebo and LO have identical shape, color, taste and weight. the doses will be administered at doses corresponding to the losartan.
  Omega-3 fish oil: The Omega-3 fish oil will be provided in 700 mg gelcaps. The starting dose will be 1.4 g/day of fish oil and continue until the 6 month visit. If the average of IL-6 measured at 3- and 6-month visits does not decrease by >40% vs. baseline (average of screening visits 1 and 2), we increase the dose to 2.8 g/day.
  Cellulose Based (Losartan Placeb
- Fish Oil Placebo + Losartan Active: This group will receive a placebo which will be matching to the Omega-3 fish oil. The placebo corn oil are obtained in gel caps and they have identical shape, color, taste and weight. The doses will be administered at doses corresponding to the Omega-3 fish oil.
  In addition, this group will receive the Losartan which will be administered at a starting dose of 25 milligrams per day. Based on tolerability, losartan will continue at a dose of either 25 milligrams /day or 50 milligrams per day for the first six months. Based on continued tolerability and inflammation level, dose may either continue at 25 or 50 milligrams per day or be increased to 100 milligrams per day for the remaining six months.
  Losartan: The Losartan will be provided in 25 mg and 50 mg capsules. The starting dose will be 25 mg/day, if tolerated, then stepped up to 50 mg/day. If there are no safety concerns, a continuation of 50 mg/day will be provided until the 6 month visit. If the average of IL-6 measure
- Total: Total of all reporting groups
Arm/Group | Fish Oil Active | Fish Oil Placebo | Losartan Active | Losartan Placebo | Fish Oil Active + Losartan Active | Fish Oil Active + Losartan Placebo | Fish Oil Placebo + Losartan Active | Fish Oil Placebo + Losartan Placebo | Total
Number analyzed (Participants) | 109 | 71 | 26 | 17 | 26 | 13 | 13 | 14 | 289
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 109 | 71 | 26 | 17 | 26 | 13 | 13 | 14 | 289
Age, Continuous [Mean (Standard Deviation); unit: years] | 78 (5) | 77 (5) | 78 (5) | 77 (6) | 77 (6) | 79 (7) | 76 (5) | 78 (5) | 78 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 37 | 15 | 12 | 14 | 6 | 6 | 4 | 152
  Male | 51 | 34 | 11 | 5 | 12 | 7 | 7 | 10 | 137
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Minority (non-white only),self-report | 24 | 14 | 9 | 3 | 4 | 3 | 3 | 4 | 64
Region of Enrollment [Number; unit: participants]
  United States | 109 | 71 | 26 | 17 | 26 | 13 | 13 | 14 | 289
IL-6 [Mean (Standard Deviation); unit: pg/ml] | 3.7 (1.5) | 4.4 (1.7) | 3.5 (1.3) | 5.7 (3.7) | 2.8 (1.6) | 3.1 (1.4) | 4.3 (1.2) | 4.2 (1.6) | 3.9 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Interleukin-6 Level Between Groups
Description: Changes in the Interleukin-6 Level Between the Groups
Time Frame: Changes from baseline to month 12
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Fish Oil Active + Losartan Active: This group will receive both the Losartan and Omega-3 fish oil. Losartan will be administered at a starting dose of 25 milligrams per day. Based on tolerability, losartan will continue at a dose of either 25 milligrams per day or 50 milligrams per day for the first six months. Based on continued tolerability and inflammation level, dose may either continue at 25 or 50 milligrams per day or be increased to 100 milligrams/day for the remaining six months.
  Omega-3 fish oil will be administered at a dose of 1.4 grams per day for the first six months. Based on tolerability and inflammation level, dose may either continue at 1.4 grams per day or be increased to 2.8 grams per day for the remaining six month.
  Omega-3 fish oil: The Omega-3 fish oil will be provided in 700 mg gelcaps. The starting dose will be 1.4 g/day of fish oil and continue until the 6 month visit. If the average of IL-6 measured at 3- and 6-month visits does not decrease by >40% vs. baseline (average of screenin
- Fish Oil Placebo + Losartan Active: This group will receive a placebo which will be matching to the Omega-3 fish oil. The placebo corn oil are obtained in gel caps and they have identical shape, color, taste and weight. The doses will be administered at doses corresponding to the Omega-3 fish oil.
  In addition, this group will receive the Losartan which will be administered at a starting dose of 25 milligrams/day. Based on tolerability, losartan will continue at a dose of either 25 milligrams per day or 50 milligrams per day for the first six months. Based on continued tolerability and inflammation level, dose may either continue at 25 or 50 milligrams per day or be increased to 100 milligrams per day for the remaining six months.
  Losartan: The Losartan will be provided in 25 mg and 50 mg capsules. The starting dose will be 25 mg/day, if tolerated, then stepped up to 50 mg/day. If there are no safety concerns, a continuation of 50 mg/day will be provided until the 6 month visit. If the average of IL-6 measure
Arm/Group | Fish Oil Active | Fish Oil Placebo | Losartan Active | Losartan Placebo | Fish Oil Active + Losartan Active | Fish Oil Active + Losartan Placebo | Fish Oil Placebo + Losartan Active | Fish Oil Placebo + Losartan Placebo
Number analyzed (Participants) | 109 | 71 | 26 | 17 | 26 | 13 | 13 | 14
pg/ml | 0 (2.4) | -0.1 (2.7) | -0.6 (1.0) | 3.8 (10.0) | -0.3 (1.0) | -0.2 (1.8) | -1.4 (0.9) | -1.0 (2.8)

2. Primary Outcome: Number of Participants Experiencing Major Mobility Disability
Description: The 400 meter walk test at usual pace is used to evaluate major mobility disability (MMD), defined as the inability to walk ¼ mile or 400 meters.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Fish Oil Active + Losartan Active: This group will receive both the Losartan and Omega-3 fish oil. Losartan will be administered at a starting dose of 25 milligrams per day. Based on tolerability, losartan will continue at a dose of either 25 milligrams per day or 50 milligrams per day for the first six months. Based on continued tolerability and inflammation level, dose may either continue at 25 or 50 milligrams/ day or be increased to 100 milligrams per day for the remaining six months.
  Omega-3 fish oil will be administered at a dose of 1.4 grams per day for the first six months. Based on tolerability and inflammation level, dose may either continue at 1.4 grams per day or be increased to 2.8 grams per day for the remaining six month.
  Omega-3 fish oil: The Omega-3 fish oil will be provided in 700 mg gelcaps. The starting dose will be 1.4 g/day of fish oil and continue until the 6 month visit. If the average of IL-6 measured at 3- and 6-month visits does not decrease by >40% vs. baseline (average of screenin
- Fish Oil Active + Losartan Placebo: This group will receive the Omega-3 fish oil which will be administered at a dose of 1.4 grams per day for the first six months. Based on tolerability and inflammation level, dose may either continue at 1.4 grams/day or be increased to 2.8 grams per day for the remaining six month.
  In addition, this group will receive a placebo which will be matching to the losartan. The placebo cellulose based capsule are obtained in 25 mg and 50 mg capsules. The shell capsules are cellulose based. Placebo and LO have identical shape, color, taste and weight. the doses will be administered at doses corresponding to the losartan.
  Omega-3 fish oil: The Omega-3 fish oil will be provided in 700 mg gelcaps. The starting dose will be 1.4 g/day of fish oil and continue until the 6 month visit. If the average of IL-6 measured at 3- and 6-month visits does not decrease by >40% vs. baseline (average of screening visits 1 and 2), we increase the dose to 2.8 g/day.
  Cellulose Based (Losartan Placeb
Arm/Group | Fish Oil Active | Fish Oil Placebo | Losartan Active | Losartan Placebo | Fish Oil Active + Losartan Active | Fish Oil Active + Losartan Placebo | Fish Oil Placebo + Losartan Active | Fish Oil Placebo + Losartan Placebo
Number analyzed (Participants) | 109 | 71 | 26 | 17 | 26 | 13 | 13 | 14
Participants | 20 | 5 | 4 | 15 | 4 | 3 | 7 | 3

3. Secondary Outcome: Short Physical Performance Battery (SPPB)
Description: A low score on the SPPB based on 4 m walk, balance & chair stands tests is a risk factor for disability, institutionalization, morbidity and mortality in initially non-disabled older persons. The summary score and components of the SPPB have good reliability (ICCs range from 0.88 to 0.92). Higher scores are better. Range 0-12.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fish Oil Active | Fish Oil Placebo | Losartan Active | Losartan Placebo | Fish Oil Active + Losartan Active | Fish Oil Active + Losartan Placebo | Fish Oil Placebo + Losartan Active | Fish Oil Placebo + Losartan Placebo
Number analyzed (Participants) | 109 | 71 | 26 | 17 | 26 | 13 | 13 | 14
units on a scale | 8.6 (2.3) | 8.1 (2.5) | 8.2 (2.5) | 8.4 (2.7) | 8.6 (2.5) | 7.3 (2.1) | 8.5 (2.1) | 9.1 (2.0)

4. Secondary Outcome: Number of Participants Exhibiting Frailty
Description: Frailty will be characterized with Fried criteria developed by Fried et al. that employ self-reported exhaustion, unintentional weight loss, low energy expenditure, slow gait speed, and weak grip strength. Those with >3 of the 5 factors are judged to be frail, those with 1 or 2 factors as pre-frail, and those with no factors as non-frail.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Fish Oil Active | Fish Oil Placebo | Losartan Active | Losartan Placebo | Fish Oil Active + Losartan Active | Fish Oil Active + Losartan Placebo | Fish Oil Placebo + Losartan Active | Fish Oil Placebo + Losartan Placebo
Number analyzed (Participants) | 109 | 71 | 26 | 17 | 26 | 13 | 13 | 14
Participants | 15 | 3 | 4 | 1 | 3 | 3 | 1 | 1

5. Secondary Outcome: Isometric Hand Grip Strength
Description: The purpose of this test is to measure the maximum isometric strength of the hand and forearm muscles. Scoring will be taken from the best results of 3 trials. Males scores range from 88 pounds as very poor to 141 pounds as excellent with an average of 105-113 pounds. Females scores range from 44 pounds as very poor to 84 pounds as excellent with an average of 57-65 pounds.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Fish Oil Active | Fish Oil Placebo | Losartan Active | Losartan Placebo | Fish Oil Active + Losartan Active | Fish Oil Active + Losartan Placebo | Fish Oil Placebo + Losartan Active | Fish Oil Placebo + Losartan Placebo
Number analyzed (Participants) | 109 | 71 | 26 | 17 | 26 | 13 | 13 | 14
pounds | 24.8 (8.5) | 25.3 (7.3) | 25.9 (9.2) | 27.5 (11.0) | 22.4 (9.5) | 19.8 (8.7) | 27.6 (8.4) | 23.6 (10.1)

6. Secondary Outcome: Peak Torque of the Knee Extensor and Flexor Muscles
Description: Peak torque was measured at a rotational speed of 60 degrees per second using a commercially-available Isokinetic Dynamometer (Biodex). Torque was measured during maximal knee extension and flexion reported in Newton Meters.
Time Frame: month 12
Measure: Mean (Standard Deviation); unit: Newton meters
Arm/Group | Fish Oil Active | Fish Oil Placebo | Losartan Active | Losartan Placebo | Fish Oil Active + Losartan Active | Fish Oil Active + Losartan Placebo | Fish Oil Placebo + Losartan Active | Fish Oil Placebo + Losartan Placebo
Number analyzed (Participants) | 109 | 71 | 26 | 17 | 26 | 13 | 13 | 14
Newton meters | 81.3 (34.0) | 77.7 (30.8) | 87.6 (35.5) | 78.6 (28.6) | 85.3 (29.8) | 76.6 (19.2) | 84.0 (52.8) | 86.1 (24.5)

7. Secondary Outcome: Short Form Health Survey (SF-36) - Physical Component Score
Description: The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Range: 0-100. A lower score indicates more disability, i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: month 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fish Oil Active | Fish Oil Placebo | Losartan Active | Losartan Placebo | Fish Oil Active + Losartan Active | Fish Oil Active + Losartan Placebo | Fish Oil Placebo + Losartan Active | Fish Oil Placebo + Losartan Placebo
Number analyzed (Participants) | 109 | 71 | 26 | 17 | 26 | 13 | 13 | 14
score on a scale | 41.9 (7.9) | 42.6 (9.7) | 41.8 (9.8) | 41.3 (9.0) | 41.9 (8.6) | 42.7 (8.2) | 46.6 (7.4) | 47.9 (6.7)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from each participant beginning with screening until closeout of the study. Participants were queried quarterly (every 3 months) but could report adverse events in-between visits. Participants were followed for 12 months.
Description: To minimize reporting bias, adverse events originating from the reported event collected during assessment visits are presented. These were completed every 3 months.
Arm/Group | Fish Oil Active | Fish Oil Placebo | Losartan Active | Losartan Placebo | Fish Oil Active + Losartan Active | Fish Oil Active + Losartan Placebo | Fish Oil Placebo + Losartan Active | Fish Oil Placebo + Losartan Placebo
All-Cause Mortality (participants affected / at risk) | 0/109 | 2/71 | 1/26 | 0/17 | 0/26 | 0/13 | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 30/109 | 17/71 | 3/26 | 4/17 | 8/26 | 3/13 | 2/13 | 5/14
Other Adverse Events (participants affected / at risk) | 73/109 | 46/71 | 22/26 | 16/17 | 20/26 | 12/13 | 10/13 | 11/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fish Oil Active (N=109) | Fish Oil Placebo (N=71) | Losartan Active (N=26) | Losartan Placebo (N=17) | Fish Oil Active + Losartan Active (N=26) | Fish Oil Active + Losartan Placebo (N=13) | Fish Oil Placebo + Losartan Active (N=13) | Fish Oil Placebo + Losartan Placebo (N=14)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — ANY SAE
AMNESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
AORTIC VALVE DISEASE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — ANY SAE
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
BRONCHIAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
CARDIAC DISORDERS - OTHER, SPECIFY (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
CHEST PAIN - CARDIAC (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
COLONIC HEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — ANY SAE
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — ANY SAE
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — ANY SAE
ESOPHAGEAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
FALL (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
HEART FAILURE (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
HEMATOMA (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
HEPATIC FAILURE (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — ANY SAE
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
INTRACRANIAL HEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — ANY SAE
JOINT RANGE OF MOTION DECREASED LUMBAR SPINE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
LUNG INFECTION (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — ANY SAE
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - OTHER, SPECIFY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — ANY SAE
ORTHOPEDIC NEUROLOGIC (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
RENAL AND URINARY DISORDERS - OTHER, SPECIFY (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — ANY SAE
RENAL CALCULI (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
SCALP PAIN (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
SICK SINUS SYNDROME (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
SINUS BRADYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
SKIN INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — ANY SAE
STROKE (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — ANY SAE
SURGICAL AND MEDICAL PROCEDURES - OTHER, SPECIFY (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) — ANY SAE
SURGICAL AND MEDICAL PROCEDURES, OTHER, LEFT KNEE REPLACEMENT (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
SYNCOPE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
TRANSIENT ISCHEMIC ATTACKS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
TREMOR (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
UPPER RESPIRATORY INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — ANY SAE
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — ANY SAE
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — DEATH
HEART FAILURE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — DEATH
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — DEATH
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — INPATIENT HOSP
AMNESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
AORTIC VALVE DISEASE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — INPATIENT HOSP
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
BRONCHIAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
CARDIAC DISORDERS - OTHER, SPECIFY (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
CHEST PAIN - CARDIAC (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
COLONIC HEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — INPATIENT HOSP
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — INPATIENT HOSP
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — INPATIENT HOSP
ESOPHAGEAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
FALL (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
HEART FAILURE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
HEMATOMA (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
HEPATIC FAILURE (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — INPATIENT HOSP
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
INTRACRANIAL HEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — INPATIENT HOSP
JOINT RANGE OF MOTION DECREASED LUMBAR SPINE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
LUNG INFECTION (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — INPATIENT HOSP
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - OTHER, SPECIFY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — INPATIENT HOSP
ORTHOPEDIC NEUROLOGIC (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
RENAL AND URINARY DISORDERS - OTHER, SPECIFY (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — INPATIENT HOSP
RENAL CALCULI (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
SCALP PAIN (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
SICK SINUS SYNDROME (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
SINUS BRADYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
SKIN INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — INPATIENT HOSP
STROKE (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — INPATIENT HOSP
SURGICAL AND MEDICAL PROCEDURES - OTHER, SPECIFY (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) — INPATIENT HOSP
SURGICAL AND MEDICAL PROCEDURES, OTHER, LEFT KNEE REPLACEMENT (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
SYNCOPE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
TRANSIENT ISCHEMIC ATTACKS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
TREMOR (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
UPPER RESPIRATORY INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — INPATIENT HOSP
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — INPATIENT HOSP
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - OTHER, SPECIFY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — OTHER SERIOUS EVENT
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fish Oil Active (N=109) | Fish Oil Placebo (N=71) | Losartan Active (N=26) | Losartan Placebo (N=17) | Fish Oil Active + Losartan Active (N=26) | Fish Oil Active + Losartan Placebo (N=13) | Fish Oil Placebo + Losartan Active (N=13) | Fish Oil Placebo + Losartan Placebo (N=14)
NON-SERIOUS AES - Any Adverse Event (General disorders) | 73 (166) | 46 (97) | 22 (74) | 16 (35) | 20 (46) | 12 (34) | 10 (21) | 11 (34) — Any Adverse Event
NON-SERIOUS AES - Atrial Fibrillation (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Atrial Fibrillation
NON-SERIOUS AES - Cough (General disorders) | 4 (4) | 3 (4) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 2 (2) — Cough
NON-SERIOUS AES - Dizziness/Presyncope (General disorders) | 1 (1) | 1 (1) | 6 (6) | 4 (4) | 5 (6) | 2 (2) | 5 (5) | 2 (3) — Dizziness/Presyncope
NON-SERIOUS AES - Fall (mechanical) (General disorders) | 10 (10) | 7 (7) | 1 (1) | 3 (4) | 2 (4) | 4 (5) | 0 (0) | 2 (3) — Fall (mechanical)
NON-SERIOUS AES - Fatigue (General disorders) | 2 (2) | 3 (4) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) — Fatigue
NON-SERIOUS AES - Syncope (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Syncope
NON-SERIOUS AES - GI Upset (General disorders) | 7 (7) | 5 (5) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 2 (2) — GI Upset
NON-SERIOUS AES - Hyperglycemia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Hyperglycemia
NON-SERIOUS AES - Hyperkalemia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Hyperkalemia
NON-SERIOUS AES - Severe Hyperglycemic Episode (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Severe Hyperglycemic Episode
NON-SERIOUS AES - Drop in hemoglobin (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Drop in hemoglobin
NON-SERIOUS AES - Hypotension (General disorders) | 6 (6) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Hypotension
NON-SERIOUS AES - Drop in eGFR (General disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 1 (1) — Drop in eGFR
NON-SERIOUS AES - Acute Renal Failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Acute Renal Failure
NON-SERIOUS AES - Angiodema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Angiodema
NON-SERIOUS AES - Stroke or TIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Stroke or TIA
NON-SERIOUS AES - Other (General disorders) | 69 (144) | 40 (80) | 20 (64) | 15 (26) | 19 (32) | 10 (27) | 7 (15) | 11 (29) — Other

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-10-18): https://cdn.clinicaltrials.gov/large-docs/66/NCT02676466/Prot_SAP_000.pdf
  • Informed Consent Form (2017-01-06): https://cdn.clinicaltrials.gov/large-docs/66/NCT02676466/ICF_001.pdf